CLINICAL TRIAL: NCT01974817
Title: Streptococcus Pneumoniae Colonization and Immunogenicity of 13-valent Conjugate Pneumococcal Vaccine in Patients 50 Years or Older With End Stage Renal Disease on Dialysis.
Brief Title: Study Response of 13-valent Conjugate Pneumococcal Vaccine in Patients With End Stage Renal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Subhashis Mitra, Assistant Professor of Medicine, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI170883
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-09

CONDITIONS: End Stage Renal Disease
Keywords: pneumococcal vaccine; end stage renal disease; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): Patients will receive one dose of 0.5 ml 13-valent conjugate pneumococcal vaccine (Prevnar-13) intra-muscularly.
  Interventions: Biological: 13-valent conjugate pneumococcal vaccine

INTERVENTIONS:
Biological: 13-valent conjugate pneumococcal vaccine — 0.5ml IM for one dose
  Other Names: Prevnar-13

SUMMARY:
The purpose of the study is to determine the response of 13-valent conjugate pneumococcal vaccine in patients 50 years or older with end stage renal disease on dialysis.

The study will also try to determine Streptococcus pneumoniae colonization in patients 50 years or older with end stage renal disease on dialysis.

DETAILED DESCRIPTION:
The purpose of the study is to determine the immunogenicity of 13-valent conjugate pneumococcal vaccine in patients 50 years or older with end stage renal disease on dialysis. Patients will receive one dose of 0.5ml of Prevnar-13 intra-muscularly. Antibody response to pneumococcal serotypes will be studied ar 2months and 12 months after administration of vaccine.

The study will try to determine Streptococcus pneumoniae colonization in patients 50 years or older with end stage renal disease on dialysis and also investigate if there are any change in Streptococcus pneumoniae colonization after Prevnar-13 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 50years of age with End stage renal disease on dialysis (both hemodialysis and peritoneal dialysis).
* Scheduled to receive pneumococcal vaccine either after 5years of previous vaccination or starting vaccination as part of standard care during the study period

Exclusion Criteria:

* History of S. pneumoniae infection within the last 5 years
* Vaccinated with an influenza- or diphtheria-containing vaccine within the last 6 months
* History of any severe adverse reaction associated with a vaccine
* Received gamma-globulins within the previous 6 months
* Known or suspected HIV or on immunosuppressive medications.
* Functional or anatomic asplenia
* serious chronic medical condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhashis Mitra, M.D, Principal Investigator — Michigan State University
Locations (1):
- Sparrow Dialysis at Saint Lawrence Campus, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitra S, Stein GE, Bhupalam S, Havlichek DH. Immunogenicity of 13-Valent Conjugate Pneumococcal Vaccine in Patients 50 Years and Older with End-Stage Renal Disease and on Dialysis. Clin Vaccine Immunol. 2016 Nov 4;23(11):884-887. doi: 10.1128/CVI.00153-16. Print 2016 Nov. PMID 27581438

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine
Started | 25
Completed | 17
Not Completed | 8
Not completed — Death | 4
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 9
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Antibody Concentrations After 13-valent Conjugate Pneumococcal Vaccination in in Patients 50 Years or Older With End Stage Renal Disease on Dialysis
Description: Study the immunologic response after administration of single dose 13-valent conjugate pneumococcal vaccine in patients 50 years or older with end stage renal disease on dialysis.
Time Frame: 12 months
Measure: Geometric Mean (95% Confidence Interval); unit: µg/ml
Groups:
- Vaccine Arm: A total of 17 patients received 1 dose of 13-valent pneumococcal conjugate vaccine.
Arm/Group | Vaccine Arm
Number analyzed (Participants) | 17
µg/ml
  Serotype 1 | 1.46 [0.80 to 2.64]
  Serotype 3 | 0.79 [0.43 to 1.46]
  Serotype 4 | 0.57 [0.37 to 0.87]
  Serotype 5 | 2.80 [1.30 to 6.01]
  Serotype 6A | 1.93 [0.86 to 4.32]
  Serotype 14 | 5.95 [3.07 to 11.52]
  Serotype 19F | 4.56 [2.90 to 7.18]
  Serotype 23F | 2.24 [1.11 to 4.52]
  Serotype 6B | 3.08 [1.49 to 6.36]
  Serotype 7F | 2.48 [1.29 to 4.77]
  Serotype 18C | 4.23 [2.48 to 7.19]
  Serotype 19A | 3.11 [1.38 to 6.99]
  Serotype 9V | 1.36 [0.88 to 2.09]

ADVERSE EVENTS:
Arm/Group | Vaccine Arm
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Arm (N=25)
Pain (General disorders) | 2 — Pain at the site of inhjection
Muscle pain (General disorders) | 2 — Muscle pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No